CLINICAL TRIAL: NCT06348472
Title: The Predictive Role of Immune-inflammatory Biomarkers and Their Interaction With the Oxytocin System in Trauma-related Psychotherapy Responsiveness
Status: Recruiting | Type: Observational
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Principal Investigator, Yuval Bloch, Professor, Shalvata Mental Health Center
Other Study IDs: 0004-24-SHA
Record Dates: First submitted 2024-03-17; First posted 2024-04-04 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Oxytocin and inflammatory biomarkers will be measured in saliva according to guidelines (Zilcha-Mano et al., 2020; Szabo & Slavish, 2021). The following inflammatory biomarkers will be assessed due to previously established associations with PTSD: IL-1β, IL-6, TNF-α, and CRP (Hori & Kim, 2019).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite a range of treatments for posttraumatic stress disorder (PTSD), only a small proportion of patients reach full symptomatic remission. Recent developments in the field of neuroscience have been providing compelling evidence to suggest that neurobiological determinants might influence not only the emergence of PTSD, but also its resistance to treatment. Immune-inflammation regulatory processes were found to be active during recovery from PTSD, potentially through interactive relationship with the oxytocin secretion system. This innovative longitudinal study aims to examine the role of inflammatory biomarkers and their interactive effect with the oxytocin (OT) system on the development of PTSD and on treatment response among patients with PTSD symptoms undergoing psychotherapy treatment. Patients (N = 100) suffering from trauma-related distress will be recruited from the trauma clinic in Shalvata Mental Health Center. Participants will be followed for 12 weeks of once-a-week psychotherapy sessions. They will be measured for endogenous OT level and cytokines levels in saliva before and after sessions 1, 6, and 12, and will complete psychotherapy outcome self-report questionnaires following each of these sessions.

ELIGIBILITY:
Inclusion Criteria:

* Minimum score of 33 on the PTSD symptoms questionnaire (PCL-5).
* Anticipated 12-24 psychotherapy sessions.

Exclusion Criteria:

* Psychotic episode.
* Female patients: pregnancy or breastfeeding (according to self-report).

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients demonstrating PTSD symptoms following a traumatic event, seeking psychotherapy treatment in Shalvata Mental Health Center's trauma clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Oxytocin Secretion | 12-16 weeks, depending on treatment duration
  Endogenous oxytocin level in saliva
Inflammatory Response: IL-1β | 12-16 weeks, depending on treatment duration
  inflammatory biomarker IL-1β assessed in saliva
Inflammatory Response: IL-6 | 12-16 weeks, depending on treatment duration
  inflammatory biomarker IL-6 assessed in saliva
Inflammatory Response: TNF-α | 12-16 weeks, depending on treatment duration
  inflammatory biomarker TNF-α assessed in saliva
Posttraumatic stress disorder symptoms | 12-16 weeks, depending on treatment duration
  PTSD checklist for DSM-5 (PCL-5): Self-report questionnaire consisting of 20 items ranging from 0-4. High scores indicate worst outcome.
Depression severity | 12-16 weeks, depending on treatment duration
  Patient health questionnaire (PHQ-9): Self-report questionnaire consisting of 9 items ranging from 0-3. High scores indicate worst outcome.
General anxiety symptoms | 12-16 weeks, depending on treatment duration
  Generalized anxiety disorder (GAD-7): Self-report questionnaire consisting of 7 items ranging from 0-3. High scores indicate worst outcome.

SECONDARY OUTCOMES:
Psychological resilience | 12-16 weeks, depending on treatment duration
  Conor-Davidson resilience scale (CD-RISC-10): Self-report questionnaire consisting of 10 items ranging from 0-4. High scores indicate better outcome.
Working Alliance | 12-16 weeks, depending on treatment duration
  Short Alliance Inventory (SAI): Self-report questionnaire consisting of 6 items ranging from 0-5. High scores indicate better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata Mental health Center, Hod HaSharon, Israel